CLINICAL TRIAL: NCT05793645
Title: Clinical Investigation to Assess the Feasibility of a New Diabetes Management Program, the dALi System, for Pediatric Type 1 Diabetes (T1D) Subjects
Brief Title: Clinical Investigation to Assess the Feasibility of a New Diabetes Management Program
Acronym: ODIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Key2Compliance (Industry); NordicInfu Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-22-002
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized care plan (Experimental): A personalized care plan will be deployed according to patient profile/ disease characteristics
  Interventions: Device: personalized care plan

INTERVENTIONS:
Device: personalized care plan — Algorithm that defines personalized care plan

SUMMARY:
The goal of this interventional study is to assess the adherence to a personalized care plan in patients (12-15 years) with Type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12-15 years of age.
* T1D diagnosis minimum 8 months prior to the Screening/Initiation visit (Visit 0).
* Equipped with Continuous Glucose Monitoring (CGM) System, intermittent or real-time, either alone or associated with an insulin pump system
* Subject and health care provider must use a Remote diabetes management platform for the upload and follow-up of CGM, pump data or HCL data (e.g.: Glooko, Diasend).
* Parent or guardian able and willing to give informed consent for the subject's participation in the investigation.

Exclusion Criteria:

* Initiation of use of HCL System during the last 2 months or during the investigation.
* Use of Medtronic insulin pump.
* Any disease or other medical condition, prior or concomitant medication /treatment

  /intervention, that may affect this clinical investigation or in other ways make the subject unsuitable for participation in this investigation, according to the judgement of the Principal Investigator (PI), or authorized designee.
* Participation in any clinical investigation or study within the previous 30 days, that may affect the safety or performance of this investigation.
* Mental incapacity precluding understanding or cooperation.
* Subject not able to read and communicate in Swedish without an interpreter.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of adherence | 15 weeks
  Percentage of patients adherent to the use of personalized care plan

SECONDARY OUTCOMES:
Evaluation of the children satisfaction with regards to the intervention | 15 weeks
  Evaluation of the children satisfaction with the intervention using a likert scale at the end of the intervention
Evaluation of the parents satisfaction with regards to the intervention | 15 weeks
  Evaluation of the parents satisfaction with the intervention using a likert scale at the end of the intervention
Change of MIND Youth-Questionnaire (MY-Q) score from the baseline phase to the post- intervention phase. | 15 weeks
  The total score is calculated as the mean of 27 items. Higher score represent better QoL.
Assessment of empowerment using Gothenburg Young Persons Empowerment Scale- Diabetes (GYPES) | 15 weeks
  GYPES is a validated 15 items likert scale questionnaire measured at baseline phase and post intervention
Change of PedsQL Diabetes module score from the baseline phase to the post- intervention phase. | 15 weeks
  The PedsQL Diabetes Module (PedsQL) is a validated 28-items likert scale questionnaire designed to assess diabetes-specific Helath Related Quality of Life children and adolescents. It contains questions related to diabetes management.
Change in the estimated HbA1c from the baseline phase and post intervention | 15 weeks
  The estimated HbA1c is based on average glucose measured continuously
Evolution of patient glycemic parameters from baseline to the end of intervention | 15 weeks
  Glycemic parameters measured are the Time in Range (TIR), the Time Above Range (TAR) and the Time Below Range (TBR). TIR, TAR and TBR refer to the percentage of CGM readings and time per day within, above and below the target glucose range
Description of Adverse events | Through study completion, an average of 15 weeks
  All adverse events recorded by the investigator during the study period

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Helsingborg Lasarett, Helsingborg
  - Sachsska, barn- och ungdomssjukhuset, Stockholm
  - Norrlands universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: Undecided